CLINICAL TRIAL: NCT05635188
Title: Impact of Surgical Technique (Laparoscopic, Open or Trephine) on Post-operative Complications in Urgency Ostomy Confection - a Single Center Retrospective Cohort
Brief Title: Impact of Surgical Technique on Post-operative Complications in Urgency Ostomy Confection
Status: Completed | Type: Observational
Sponsor: Instituto do Cancer do Estado de São Paulo (Other)
Responsible Party: Principal Investigator, Gabriella Rosceli Campos Zerbetto, Principal Investigator, Instituto do Cancer do Estado de São Paulo
Other Study IDs: 4.834.729
Record Dates: First submitted 2022-11-22; First posted 2022-12-02 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-12

CONDITIONS: Colostomy Stoma; Colostomy Complication; Obstruction Bowel; Surgical Complication; Surgical Procedure, Unspecified
Keywords: colostomy; laparoscopy; ostomy
MeSH Terms: conditions — Intestinal Obstruction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Open Surgery
  Interventions: Procedure: Intestinal ostomy confection
- Laparoscopic Surgery
  Interventions: Procedure: Intestinal ostomy confection
- Trephine Surgery
  Interventions: Procedure: Intestinal ostomy confection

INTERVENTIONS:
Procedure: Intestinal ostomy confection — Surgical procedure for fecal diverting

SUMMARY:
This is a single-center retrospective cohort study on cancer patients who underwent emergency ostomy. Our objective was to compare the incidence of surgical complications as well as the length of hospital stay among three different techniques for ostomy confection (laparotomy, the conventional local approach, described as trephination, and laparoscopy).

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent emergency colostomy or ileostomy

Exclusion Criteria:

* Patients who underwent other major procedures at the time of the surgery, such as enterectomy, colectomy, or tumor or other organ resection

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who underwent emergency surgery between 2008 and 2019 by the surgical team of the Cancer Institute of São Paulo State (Instituto do Câncer do Estado de São Paulo - ICESP)
Sampling Method: Non-Probability Sample
Enrollment: 154 (Actual)
Dates: Start 2008-01 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
Surgical complications | Between cohort enter (2008-2019) and study finish (2021)
  Early and late surgical complications related to the stoma and severe complications

SECONDARY OUTCOMES:
Postoperative length of hospital stay | Between cohort enter (2008-2019) and study finish (2021)
  Length of hospital stay after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Gabriella Rosceli C Zerbetto, Principal Investigator — Instituto do Cancer do Estado de São Paulo
Locations (1):
- Instituto do Câncer do Estado de São Paulo - ICESP, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
We intend to publish the results of the study, but not make available individual participant date